CLINICAL TRIAL: NCT05112172
Title: The Impact of Hypoxia on Patients With Precapillary Pulmonary Hypertension and Treatment of Adverse Effects
Brief Title: Effect of Oxygen Therapy for Patients With Precapillary Pulmonary Hypertension Who Experience an Altitude Related Adverse Health Effect (ARAHE) During 30h Exposure to 2500m
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OVERALP II B
Record Dates: First submitted 2021-10-14; First posted 2021-11-08 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: High Altitude Pulmonary Hypertension; Oxygen Therapy
MeSH Terms: conditions — Pulmonary edema of mountaineers | interventions — Oxygen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxygen Therapy (Experimental): Oxygen Therapy in patients developing an altitude related adverse health effect (ARAHE) during 30h exposure to 2500m of high altitude
  Interventions: Other: Oxygen Therapy

INTERVENTIONS:
Other: Oxygen Therapy — Oxygen Therapy in patients developing an altitude related adverse health effect (ARAHE) during 30h exposure to 2500m of high altitude

SUMMARY:
To study whether oxygen therapy titrated to maintain oxygenation (SpO2) > 90% at 2500m would resolve altitude-related adverse health effects, symptoms and impaired exercise during 30h exposure to high altitude.

DETAILED DESCRIPTION:
Patients with pulmonary hypertension who reveal an altitude-related adverse health effects at 2500m will be given oxygen therapy by nasal cannula titrated to maintain the oxygen saturation above 90%. The study will investigate, whether this measure will restore altitude-induced impairment to baseline levels at low altitude.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* PH class I (PAH) or IV (CTEPH) diagnosed according to guidelines: mean pulmonary artery pressure >20 mmHg, pulmonary vascular resistance ≥3 wood units, pulmonary arterial wedge pressure ≤15 mmHg during baseline measures at the diagnostic right-heart catheterization

Exclusion Criteria:

* resting partial pressure of oxygen <8 kilopascal at Zurich at 490 m low altitude
* exposure to an altitude >1000 m for ≥3 nights during the last 2 weeks before the study
* inability to follow the procedures of the study
* other clinically significant concomitant end-stage disease (e.g., renal failure, hepatic dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Recovery from ARAHE | 30 hours
  Proportion of patients with precapillary pulmonary hypertension experiencing an ARAHE at 2500 m of high altitude and receiving oxygen therapy titrated to achieve SpO2 ≥ 90% who recover from ARAHE, have improved symptoms and achieve constant work-rate exercise time within a minimal important difference as defined for patients with respiratory disease within 1.75 min of baseline value at 490 m; time frame within 6 h after initiation of oxygen therapy.

SECONDARY OUTCOMES:
Constant work-rate exercise time | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude in constant work-rate exercise time cycle exercise test at 75% Wmax at low altitude
Maximum work-rate in incremental ramp cycle exercise tests | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude in maximal exercise capacity during a incremental ramp cycle exercise test
Hemodynamics | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude in hemodynamics assessed by echocardiography at rest including pulmonary artery pressure, cardiac output, pulmonary vascular resistance and right heart function assessed as tricuspid plane systolic excursion and fractional area change.
Borg dyspnoea scale | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude baseline in post-exercise Borg dyspnoea scale going from 1-10 scores with higher values meaning worse dyspnea
Visual Analogue Scale | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude baseline in symptoms assessed by the Visual Analogue Scale for dyspnoea, a 10cm line from left to right where patients have to add a cross-line with higher values meaning better feeling.
Cognitive testing | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude baseline in cognitive function tests
sit-to-stand test | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude baseline in sit-to-stand test
Sleep disordered breathing | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude in sleep disordered breathing
6 minute walk test | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude in 6 minute walk test
Acute Mountain Sickness Score | 30 hours
  Difference with oxygen therapy at high altitude vs. low altitude baseline in symptoms assessed by the Lake Louise acute mountain sickness score going from 0-12 points with mild AMS as 3-5 points, moderate AMS as 6-9 points, and severe AMS as 10-12 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland